CLINICAL TRIAL: NCT04426071
Title: COVID-19 and Disability: The Impact of a Societal Lockdown on Those With Spinal Cord and Brain Injuries
Brief Title: The Impact of a Societal Lockdown on Those With Spinal Cord and Brain Injuries
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 115999
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Brain Injuries; Stroke; Spinal Cord Injuries
Keywords: Stroke; Spinal Cord Injury; Brain Injury; COVID; Access to health care; Mental Health
MeSH Terms: conditions — Brain Injuries; Stroke; Spinal Cord Injuries; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCI, brain injury, stroke Participants: Those 18 years of age and older, diagnosed with a stroke, spinal cord injury (traumatic and non-traumatic), or acquired brain injury (of all severities, including concussion) living in the community will be included. Additionally, only those the cognitive capacity to understand and complete the measures will be included. Those who consent will complete an online survey on enrollment into the study, and subsequently at 3 and 6 months.

SUMMARY:
Document and evaluate the impact of societal restrictions due to the pandemic on SCI- and ABI-related disability and functional impairments, and the resultant effects on psychological wellbeing, physical wellbeing and quality of life for those with SCI/ABI.

DETAILED DESCRIPTION:
The investigators will conduct a longitudinal survey to examine the impact of COVID19 on those with SCI and ABI. An a priori sample size of 117 individuals based on an alpha level of .05 and level of acceptable error at 3% was calculated. Anticipating for loss to follow up rate of up to 20%, a total of 142 participants will be recruited. Patients will be recruited among those who attend virtual medical appointments at Parkwood Institute for ABI and SCI. We will also liaise with SCI-Ontario and the Ontario Brain Injury Association to assist in the recruitment of additional participants. Those who consent will complete an online survey on enrollment into the study, and subsequently at 3 and 6 months. Demographic data of the individuals participating in the study will be recorded. Participants' access to health care services will be evaluated using the following subdomains: medical care, complementary care, medications/equipment, satisfaction/acceptability, affordability, ability to engage, and indirect support.

ELIGIBILITY:
Inclusion Criteria:

* stroke, spinal cord injury (traumatic and non-traumatic) or acquired brain injury (of all severities, including concussion)
* live in the community
* have the cognitive capacity to understand and complete the measures

Exclusion Criteria:

* does not have the cognitive capacity to understand and complete the measures
* does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those 18 years of age and older with stroke, spinal cord injury (traumatic and non-traumatic) or acquired brain injury (of all severities, including concussion) living in the community will be included. Additionally, only those the cognitive capacity to understand and complete the measures will be included.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fear of COVID-19 | baseline, 3 months, 6 months
  Fear of COVID-19 Questionnaire

SECONDARY OUTCOMES:
Change in ability to participate in social roles and activities | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Ability to Part. in SRA
Change in depressive symptoms | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Depression
Change in positive affect and well-being | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Pos. Affect & Well-Being
Change in anxiety | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Anxiety
Change in fatigue | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Fatigue
Change in emotional and behavioural dyscontrol | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Emotional & Beh. Dyscontrol
Change in satisfaction with social roles and activities | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Satisfaction w SRA
Change in sleep disturbance | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Sleep Disturbance
Change in stigma | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Stigma
Change in cognitive function | baseline, 3 months, 6 months
  NeuroQol SF v1.0 - Cognitive Function
Change in social distancing strategies used | baseline, 3 months, 6 months
  23 questions about strategies to social distance
Change in thoughts and feelings about social distancing | baseline, 3 months, 6 months
  22 questions about social distancing

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Loh, MD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada